CLINICAL TRIAL: NCT01833520
Title: Phase I Dose Escalation of Monthly Intravenous Ra-223 Dichloride in Osteosarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0952; NCI-2013-02267 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Sarcoma
Keywords: Sarcoma; Osteosarcoma; recurrent or metastatic; Ra-223 dichloride; Radium-223 chloride; Alpharadin
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ra-223 Dichloride (Experimental): Phase I Starting Dose of Ra-223 Dichloride: 50 kBq/kg by vein over several minutes on Day 1 of each 4-week cycle.
  Phase II Starting Dose of Ra-223 Dichloride: MTD from Phase I.
  Up to 3 groups of 3 participants will be enrolled in the Phase I portion of the study, and up to 6 participants will be enrolled in Phase II.
  Interventions: Drug: Ra-223 Dichloride

INTERVENTIONS:
Drug: Ra-223 Dichloride — Phase I Starting Dose of Ra-223 Dichloride: 50 kBq/kg by vein over several minutes on Day 1 of each 4-week cycle.
  Phase II Starting Dose of Ra-223 Dichloride: MTD from Phase I.
  Other Names: Alpharadin

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of radium-223 dichloride that can be given to patients with osteosarcoma.

Radium-223 chloride is designed to work like radiation therapy in cells that are actively making bone. It is designed to target new bone growth in and around bone cancer and may kill cancer cells.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of 3 participants will be enrolled in the Phase I portion of the study, and up to 6 participants will be enrolled in Phase II.

If you are found to be eligible to take part in this study, you will be assigned to a dose level of radium-223 dichloride based on when you join this study. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of radium-223 dichloride is found.

If you are enrolled in the Phase II portion, you will receive radium-223 dichloride at the highest dose that was tolerated in the Phase I portion.

Study Drug Administration:

You will receive radium-223 chloride by vein over several minutes on Day 1 of each 4-week cycle.

You should drink plenty of fluids before each study drug dose.

You and your caregivers will receive spoken and written instructions about safety precautions after receiving this drug.

Study Visits:

At all study visits, you will be asked about any drugs you may be taking and if you have had any side effects from them.

On Day 1 of Cycle 2-6:

* You will have a physical exam, including measurement of your vital signs
* You will complete a brief questionnaire about any pain that you may be experiencing. This questionnaire should take about 5-10 minutes to complete.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If you can become pregnant, you will have a urine or blood pregnancy test. If the doctor thinks it is needed, you will also have an ultrasound to check for pregnancy. To take part in this study, you cannot be pregnant.

Within 1-3 weeks after Cycle 3:

* You will have scans such as a bone scan and CT or MRI scan to check the status of the disease.
* Blood (about 1 tablespoon) will be drawn for routine tests.

You may have other routine tests done, including a pregnancy test, if the study doctor thinks it is needed.

Length of Study Drug Dosing:

You may continue taking the study drug for up to 6 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in this study will be over once you have completed the end-of-dosing visit (and follow-up visits if applicable).

End-of-Dosing Visit:

About 30 days after your last study drug dose:

* You will be asked about any drugs you may be taking and if you have had any side effects from them.
* You will have a physical exam, including measurement of your vital signs.
* You will complete a brief questionnaire about any pain that you may be experiencing. This questionnaire should take about 5-10 minutes to complete.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have scans such as a bone scan and CT or MRI scan to check the status of the disease.

Follow-Up Visits:

If you are younger than 18 years old, your height and weight will be measured 1 time a year until you turn 21. These measurements may stop earlier if your height stays about the same for 2 years in a row.

Information about your health status and any side effects (especially related to your bones) will be collected and reported to the study staff every year.

This is an investigational study. Radium-223 dichloride is commercially available and FDA approved for the treatment of certain types of prostate cancer. It is currently being used for research purposes only.

Up to 20 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with progressive, locally recurrent, or metastatic osteosarcoma (i.e. high-risk only) with no standard curative options available with at least one indicator lesion avid on 99mTc-MDP scan or a Sodium Fluoride (Na F) Bone PET scan will be eligible. In addition, subjects with extremely rare bone forming osteosarcoma-like tumors that behave like osteosarcoma phenotypically and are clinically treated like osteosarcoma (eg. Malignant Fibrous Histiocytoma of Bone or malignant transformation of giant cell tumor of bone) may be included if they satisfy all of the inclusion criteria.
2. Anatomic imaging (CT or MRI) of all sites of disease along with chest CT at baseline and restaging for all patients will be done to allow for assessment of RECIST progression. RECIST progression will determine progressive disease regardless of other imaging.
3. Indicator lesion that has uptake of 99mTc-MDP on bone scan or a Sodium Fluoride ( Na F) Bone PET scan and can be subjected to quantitative assessment by this scans and possibly other means.
4. Age 15 and above and >40 kg.
5. ECOG=2 or better
6. Subjects or their guardians must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
7. All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF).
8. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
9. Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 30 days after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
10. Acceptable hematology and serum biochemistry screening values: White Blood Cell Count (WBC) >= 1500/mm3; Absolute Neutrophil Count (ANC) >= 1,000/mm3; Platelet (PLT) count >= 75,000/mm3; Hemoglobin (HGB) >= 8 g/dl; Total bilirubin level <= 1.5 x institutional upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 x ULN; Creatinine <= 1.5 x ULN; Albumin > 25 g/L
11. Willing and able to comply with the protocol, including follow-up visits and examinations.
12. Patients with progressive, locally recurrent, or metastatic osteosarcoma (i.e. high-risk only) with at least one indicator lesion avid on 99mTc-MDP scan will be eligible.

Exclusion Criteria:

1. Diagnosis other than osteosarcoma.
2. 99mTc-MDP bone scan with no significant uptake (i.e. "nothing" for a bone-seeking isotope to target/ i.e. indicator lesion that would be expected to have the bone-seeking targeted uptake of 223-radium dichloride).
3. Other malignancy treated within the last 3 years (except non-melanoma skin cancer or low-grade superficial bladder cancer).
4. Any other serious illness or medical condition, such as but not limited to: Any active infection >= National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade 2; Cardiac failure New York Heart Association (NYHA) III or IV; Fecal incontinence (this is because of Ra-223 elimination in feces).
5. Women who are pregnant or breast-feeding.
6. Inability to comply with the protocol and/or not willing or not available for follow-up assessments.
7. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
8. Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization)
9. Patients on oxygen

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Subbiah, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Subbiah V, Anderson P, Rohren E. Alpha Emitter Radium 223 in High-Risk Osteosarcoma: First Clinical Evidence of Response and Blood-Brain Barrier Penetration. JAMA Oncol. 2015 May;1(2):253-5. doi: 10.1001/jamaoncol.2014.289. No abstract available. PMID 26181034
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: October 2013 to October 2015
Groups:
- Escalation 50 kBq/kg; Escalation 75 kBq/kg; Escalation 100 kBq/kg; Expansion 100 kBq/kg: Radium-223 dichloride will be given monthly for up to 6 cycles and side effects of this bone-targeted therapy on monthly blood counts and alkaline phosphatase will be determined.
  Ra-223 dichloride will be administered as a slow bolus IV injection at intervals of every 4 weeks for up to 6 cycles.
Period: Overall Study
Arm/Group | Escalation 50 kBq/kg | Escalation 75 kBq/kg | Escalation 100 kBq/kg | Expansion 100 kBq/kg
Started | 3 | 3 | 9 | 3
Completed | 0 | 0 | 1 | 0
Not Completed | 3 | 3 | 8 | 3
Not completed — Lack of Efficacy | 3 | 3 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Escalation: Dose level: 50 kBq/kg, 75 kBq/kg and 100 kBq/kg. Radium-223 dichloride will be given monthly for up to 6 cycles and side effects of this bone-targeted therapy on monthly blood counts and alkaline phosphatase will be determined.
  Ra-223 dichloride will be administered as a slow bolus IV injection at intervals of every 4 weeks for up to 6 cycles.
- Expansion: Dose level: 100 kBq/kg. Radium-223 dichloride will be given monthly for up to 6 cycles and side effects of this bone-targeted therapy on monthly blood counts and alkaline phosphatase will be determined.
  Ra-223 dichloride will be administered as a slow bolus IV injection at intervals of every 4 weeks for up to 6 cycles.
- Total: Total of all reporting groups
Arm/Group | Escalation | Expansion | Total
Number analyzed (Participants) | 15 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 1 | 6
  Between 18 and 65 years | 9 | 2 | 11
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 13 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 12 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 3 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Ra-223 Dichloride in Osteosarcoma
Description: The goal of this initial study is to determine the safety of escalating doses of monthly Ra-223 dichloride in the number of osteosarcoma participants with osteoblastic bone-forming metastases until MTD or a dose 100 kBq/kg dose is reached (whichever is first).
Time Frame: 3 months
Measure: Number; unit: kBq/kg
Arm/Group | Escalation 100 kBq/kg | Expansion 100 kBq/kg
Number analyzed (Participants) | 9 | 3
kBq/kg | 100 | 100

2. Secondary Outcome: Number of Participants With Objective Response of Osteosarcoma Indicator Lesions to 223-Radium Dichloride
Description: Alkaline phosphatase reduction to quantitative imaging techniques (99mTc-MDP, 18FDG-PET-CT, 18FNa PET-CT scans) to determine objective response of osteosarcoma indicator lesions to 223-radium dichloride. >30% increase in SUV peak indicates progression, if >30% decrease in SUV peak indicates a response and other does not meet above criteria or mixed response using the NAFCIST and PERCIST criteria.
Time Frame: Baseline, 3 months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation 50 kBq/kg | Escalation 75 kBq/kg | Escalation 100 kBq/kg | Expansion 100 kBq/kg
Number analyzed (Participants) | 2 | 3 | 6 | 3
Participants
  >30% increase in SUV peak | 2 | 0 | 3 | 2
  >30% decrease in SUV peak | 0 | 0 | 1 | 0
  Other/Mixed Response | 0 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Escalation 50 kBq/kg | Escalation 75 kBq/kg | Escalation 100 kBq/kg | Expansion 100 kBq/kg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 5/9 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/9 | 3/3
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 4/9 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation 50 kBq/kg (N=3) | Escalation 75 kBq/kg (N=3) | Escalation 100 kBq/kg (N=9) | Expansion 100 kBq/kg (N=3)
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Neck pain (General disorders) | 0 | 0 | 1 | 0
Bronchopulmonary hemorhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Abdominal pain (General disorders) | 0 | 0 | 1 | 0
Thromboembolic event (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 0
Tumor pain (General disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alkaline phophatase increased (Endocrine disorders) | 0 | 0 | 0 | 1
Pain in extremity (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation 50 kBq/kg (N=3) | Escalation 75 kBq/kg (N=3) | Escalation 100 kBq/kg (N=9) | Expansion 100 kBq/kg (N=3)
Brittle nails (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Intermittent pain (jaw, neck, trunk, back) (General disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
White Blood Cell decreased (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0
Bone pain (General disorders) | 0 | 0 | 2 | 0
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT01833520/Prot_SAP_000.pdf